CLINICAL TRIAL: NCT02267018
Title: Effect of Nasal Continuous Positive Airway Pressure (nCPAP) Versus Non-Invasive High Frequency Ventilation (NIHFV) on the Diaphragm Electrical Activity in Very Low Birth Weight Preterm Infants
Brief Title: Diaphragm Electrical Activity of Preterm Infants on nCPAP Versus NIHFV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Michael Dunn, Staff Neonatologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 001-2014
Record Dates: First submitted 2014-10-07; First posted 2014-10-17 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: nCPAP; High-Frequency Oscillator Ventilation; Diaphragm Electrical Activity
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nCPAP (Active Comparator): Nasal continuous positive airway pressure is a frequently used modality for non-invasive respiratory support in preterm infants.
  Interventions: Device: Drager VN500 Ventilator
- NIHFV (Active Comparator): Non-invasive high-frequency ventilation is a relatively new modality that is being utilized to support preterm infants and prevent the need for invasive ventilation, but this particular modality is has not been well studied to date.
  Interventions: Device: Drager VN500 Ventilator

INTERVENTIONS:
Device: Drager VN500 Ventilator — This ventilator is capable of providing both nCPAP and NIHFV support.

SUMMARY:
Preterm babies have immature lungs and frequent pauses in their breathing which often necessitates breathing support. Nasal Continuous Positive Airway Pressure (nCPAP) is one of the most commonly used tools, but does not always provide enough support. A new option is non-invasive high frequency ventilation (NIHFV), which gently shakes the lungs to help with gas exchange and may decrease a baby's work of breathing. The investigators plan to study very low birth weight preterm babies who are generally well but require some support with their breathing. By inserting a special feeding tube with sensors into the stomach, the investigators can measure the electrical activity of the diaphragm (EAdi), which is an important muscle for breathing. By analyzing EAdi in babies receiving either nCPAP or NIHFV, the investigators will be able to measure and compare how each method of support affects a baby's breathing. This important study will help us determine the most appropriate breathing support for preterm babies.

DETAILED DESCRIPTION:
Continuous Positive Airway Pressure is one of the most researched and accepted methods of delivering NIV to term and preterm infants. Non-invasive high frequency ventilation is a relatively new method of delivering NIV respiratory support in preterm infants. Preliminary studies suggest superiority over CPAP, and NIHFV is being increasingly utilized in clinical practice in an attempt to prevent intubation and minimize ventilation-induced lung injury in preterm infants. However, little is known about its mechanism of action and its effect on respiratory mechanics in the newborn. The objective of this study is to compare the effects of non-invasive ventilation (NIV) delivered by nasal Continuous Positive Airway Pressure (nCPAP) versus Non-Invasive High Frequency Ventilation (NIHFV) on respiratory pattern as assessed by the electrical activity of the diaphragm (EAdi) in very low birth weight (VLBW) preterm infants.

We hypothesize that in VLBW preterm infants with relative pulmonary insufficiency, NIHFV will reduce respiratory drive and improve ventilation, subsequently resulting in decreased patient diaphragm energy expenditure. This would be demonstrated by decreased neural respiratory rates and/or decreased peak electrical activity of the diaphragm while breathing on NIHFV compared to nCPAP.

Clinicians are seeking alternative methods for providing non-invasive respiratory support to preterm infants. NIHFV is a relatively new modality that is being increasingly utilized in clinical practice but has not been well studied. This study will help us determine how non-invasive high frequency ventilation (NIHFV) affects breathing in preterm infants, as compared to the more traditional modality of nasal CPAP. Therefore, clinicians will not only be able to better understand how NIHFV works, but also utilize this information to decide on the most appropriate respiratory support modality for preterm patients

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable preterm infants with birth weights ≤1500g admitted to the neonatal intensive care unit (NICU) at Sunnybrook Health Sciences Centre or BC Women's and Children's Hospital.
* Patient's on nasal continuous positive airway pressure of 6 to 8 cmH20 support for at least 48 hours, treated with methylxanthines for apnea of prematurity and requiring 25-40% of oxygen.

Exclusion Criteria:

* infants with congenital anomalies of the gastrointestinal tract, phrenic nerve damage, diaphragmatic paralysis, esophageal perforation;
* infants with congenital or acquired neurological deficit (including significant intraventricular hemorrhage >Grade II) [27], neonatal seizure;
* infants with significant congenital heart disease (including symptomatic PDA);
* infant with congenital anomalies of the diaphragm;
* infant with congenital anomalies of the respiratory tracts (e.g. Congenital Cystic Adenomatoid Malformation (CCAM)) infants requiring ongoing treatment for sepsis, necrotizing enterocolitis (NEC), antibiotics for lung infections, narcotic analgesics, or gastric motility agents will be excluded.
* infants on nasal CPAP and requiring more than 40% oxygen will be excluded from the study.
* infants with significant gastric residuals and vomiting, infants with facial anomalies, infants with pneumothorax or pneumomediastinum, and infants in the immediate postoperative period will be excluded.

Ages: 2 Days to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the difference in the peak electrical activity of the diaphragm between nCPAP and NIHFV. | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (nCPAP and NIHFV).

SECONDARY OUTCOMES:
Difference in neural respiratory rate. | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (nCPAP and NIHFV).
Difference in neural inspiratory time. | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (nCPAP and NIHFV).
Difference in diaphragm energy expenditure. | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (nCPAP and NIHFV).
Difference in transcutaneous pCO2. | 4 hours
  As read from transcutaneous pCO2 monitor
Number of apnea episodes. | 4 hours
  Pauses in electrical activity of the diaphragm of greater than 5 seconds and greater than 15 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunn, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No